CLINICAL TRIAL: NCT05347537
Title: Effects of Mulligan's Mobilization With and Without Clamshell Exercise on Pain, Disability and Quality of Life in Patients With Sacroiliac Joint Dysfunction
Brief Title: Effects of Mulligan's Mobilization With and Without Clamshell Exercises in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0114 Rahat
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Sacroiliac Joint Somatic Dysfunction; Pain; Disability Physical; Treatment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan mobilization (Experimental): Group A will be treated with only mulligan's mobilization with movement at the frequency of 3 sets with 10 repetitions 3 times/ week without the clamshell exercise.
  Interventions: Other: Mulligan mobilization
- Mulligan mobilization with clamshell exercise (Active Comparator): Group B will be treated with mulligan's mobilization with movement and clamshell exercises.
  Interventions: Other: clamshell exercise

INTERVENTIONS:
Other: Mulligan mobilization — Mulligan Mobilization designed to reduce pain and improve the patient's range of motion. Mulligan's mobilization with movement at the frequency of 3 sets with 10 repetitions 3 times/ week without the clamshell exercise.
  Arms: Mulligan mobilization
Other: clamshell exercise — As a general exercise, the clamshell can help strengthen your medial glutes, bringing more power and stability to your hips. This group treated with mulligan's mobilization with movement and clamshell exercises.
  Arms: Mulligan mobilization with clamshell exercise

SUMMARY:
Sacroiliac joint dysfunction is the changing of joint structure (ligaments, muscles and cartilage) that cause impairments and movement restrictions. It is one of the primary sources of low back pain among female population and often misdiagnosed. Almost 15-30% patients are suffering from sacroiliac joint dysfunction who presented with the complaint of low back pain. The aim of the study is to determine the effect of mulligan's mobilization with and without clamshell exercise on pain, disability and quality of life in patients with sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
A Randomized controlled trial will be conducted at Fatima Memorial Hospital Physiotherapy Clinic & Boston Physiotherapy and wellness Clinic through consecutive sampling technique on 32 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A & group B. Group A will be treated with only mulligan's mobilization with movement at the frequency of 3 sets with 10 repetitions 3 times/ week without the clamshell exercise. Group B will be treated with mulligan's mobilization with movement and clamshell exercises. Outcome measures will be conducted through pain, disability and quality of life questionnaire after 6 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between the ages of 20 to 50 years with positive Leslett's criteria.
* Sacroiliac pain of sub-acute level with the duration of 4 weeks

Exclusion Criteria:

* Spondylosis
* Lumbar canal stenosis
* Spondylolisthesis
* Pervious spinal surgery
* Congenital postural deformities and
* Lumbar disc herniation
* Pelvic bone fractures

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
1. NPRS | follow up at 6th week
  Patient level of pain was assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain"
2. Oswestry Disability index (NDI) | follow up at 6th week
  It comprises 10 items, 7 related with daily activities, 2 related to pain , 1 related to concentration. Each item scores from 0 to 5. Total score is expressed as percentage with higher scores related to greater disability.
Euro Quality of life (EQ-5D) | follow up at 6th week
  Quality of life will be checked by Euro Quality of life (EQ-5D) Health Related Quality of Life Question.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphill, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Fatima memorial hospital - Physical therapy clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Added MAN, de Freitas DG, Kasawara KT, Martin RL, Fukuda TY. STRENGTHENING THE GLUTEUS MAXIMUS IN SUBJECTS WITH SACROILIAC DYSFUNCTION. Int J Sports Phys Ther. 2018 Feb;13(1):114-120. PMID 29484248
- [Background] Ramirez C, Sanchez L, Oliveira B. Prevalence of sacroiliac joint dysfunction and sacroiliac pain provocation tests in people with low back pain. Annals of Physical and Rehabilitation Medicine. 2018;61:e152.
- [Background] Sarkar M, Goyal M, Samuel AJ. Comparing the Effectiveness of the Muscle Energy Technique and Kinesiotaping in Mechanical Sacroiliac Joint Dysfunction: A Non-blinded, Two-Group, Pretest-Posttest Randomized Clinical Trial Protocol. Asian Spine J. 2021 Feb;15(1):54-63. doi: 10.31616/asj.2019.0300. Epub 2020 Jan 30. PMID 31992024
- [Background] Bashir MS, Noor R, Hadian MR, Olyaei G. Pattern of changes in latissimus dorsi, gluteus maximus, internal oblique and transverse abdominus muscle thickness among individuals with sacroiliac joint dysfunction. Pak J Med Sci. 2019;35(3):818-823. doi: 10.12669/pjms.35.3.62. PMID 31258601
- [Background] Jeong S-G, Cynn H-S, Lee J-H, Choi S, Kim D. Effect of modified clamshell exercise on gluteus medius, quadratus lumborum and anterior hip flexor in participants with gluteus medius weakness. Journal of the Korean Society of Physical Medicine. 2019;14(2):9-19.
- [Background] Ribeiro S, Heggannavar A, Metgud S. Effect of mulligans mobilization versus manipulation, along with mulligans taping in anterior innominate dysfunction-A randomized clinical trial. Indian Journal of Physical Therapy and Research. 2019;1(1):17.
- [Background] Kaur H, Sharma M, Hazari A. Effectiveness of Maitland Mobilization and Mulligan Mobilization in Sacroiliac Joint Dysfunction: A Comparative Study. Critical Reviews™ in Physical and Rehabilitation Medicine. 2019;31(2).
- [Background] Sanika V, Prem V, Karvannan H. Comparison of Glutues Maximus Activation to Flexion Bias Exercises Along with MET Technique in Subjects with Anterior Rotated Sacroiliac Joint Dysfunction-a Randomised Controlled Trial. Int J Ther Massage Bodywork. 2021 Mar 1;14(1):30-38. eCollection 2021 Mar. PMID 33654504
- [Background] Javadov A, Ketenci A, Aksoy C. The Efficiency of Manual Therapy and Sacroiliac and Lumbar Exercises in Patients with Sacroiliac Joint Dysfunction Syndrome. Pain Physician. 2021 May;24(3):223-233. PMID 33988941
- [Background] Saleh HM, Ibrahim AH, Yosef AO, Sedhom MG. EFFECT OF RADIAL EXTRA CORPOREAL SHOCK WAVE THERAPY VERSUS MULLIGAN MOBILIZATION ON SACROILIAC JOINT DYSFUNCTION. Journal of Critical Reviews. 2020;7(19):8055-9.